CLINICAL TRIAL: NCT04835194
Title: Clinical Phenotypes of Heart Failure With Preserved Ejection Fraction and Its Association With Cardiovascular Outcomes in Patients With Hypertension and Diabetes
Brief Title: Phenotypes and Outcomes of Heart Failure With Preserved Ejection Fraction in Patients With Hypertension and Diabetes
Status: Completed | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Van Ngoc-Thanh Nguyen, Principle investigator: Van Ngoc-Thanh Nguyen, MD, MSci, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: 2129-ĐHYD
Record Dates: First submitted 2021-04-03; First posted 2021-04-08 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Diabetes Mellitus, Type 2; Hypertension
Keywords: Heart failure with preserved ejection fraction; Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phenotype 1 (from LCA)
- Phenotype 2 (from LCA)
- Phenotype 3 (from LCA)

SUMMARY:
Our study is the first multicenter study in Vietnam on clinical phenotypes of heart failure with preserved ejection fraction (HFpEF) in patients with concurrent type 2 diabetes (T2DM) and hypertension (HTN). The purpose of this study is to identify different phenotypes of the Vietnamese HFpEF-HTN-T2DM population, as well as the association of these phenotypes with long-term outcomes.

DETAILED DESCRIPTION:
The study is expected to provide further understanding on the characteristics, risk profiles and treatment patterns of an emergingly common and high-risk population. At baseline, patients will be grouped into phenotypes. During the 12 month follow up, investigators will collect information on predefined outcomes, especially the all cause mortality and hospitalization for heart failure, thereby establishing the association between phenotypes and outcomes.

The knowledge gained from the study is supposed to add valuable information on the feasibility of phenotype-guided approach for heart failure with preserved ejection fraction in patients with hypertension and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years at screening
* Preexisting or newly diagnosed hypertension, diabetes
* Preexisting or newly diagnosed heart failure with preserved ejection fraction using 2016 European Society of Cardiology's guideline on heart failure.

  * Signs and symptoms of heart failure
  * N-terminal pro brain natriuretic peptide (NT-proBNP) ≥300 in acute setting, and ≥125 in chronic setting
  * Echocardiography with left ventricular ejection fraction (LVEF) ≥50% and at least one of these following criteria:

    * Structural changes indicated by either left ventricle (LV) hypertrophy (any of the following: intraventricular septal or posterior wall thickness ≥1.1 cm, and/or LV mass index ≥115 g/m*2 in male and ≥95 g/m*2 in female), or left atrium (LA) enlargement (any of the following: left atrial volume (LAV) index ≥34 ml/m*2, or or LA diameter >40 mm)
* Further inclusion criteria apply

Exclusion Criteria:

* Listed for heart transplant
* Primary stage D valvular heart disease requiring surgery or intervention, prosthetic or mechanical valve.
* Severe, unrepaired pericardiac disease
* Complex, unrepaired congenital heart disease
* Takotsubo disease, peripartum cardiomyopathy, chemotherapy-induced cardiomyopathy, cardiac sarcoidosis/amyloidosis.
* End stage renal dysfunction, defined as persistent estimated glomerular filtration rate (eGFR)<15 ml/min (CKD-EPI Chronic Kidney Disease Epidemiology Collaboration Equation) or requiring renal replacement therapy.
* Child-Pugh-Turcotte C.
* Life expectancy <1 year due to non-cardiac etiology, as per investigator judgement
* Severe pulmonary disease requiring continuous home oxygen
* Pregnancy or lactation.
* Concurrent enrolment in another interventional device or drug trial
* Further exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the outpatient clinic and/or hospital ward in two tertiary hospitals (University Medical Center, Nhan Dan Gia Dinh hospital) and one heart center (Heart Institute in Ho Chi Minh city).
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Phenotypes of heart failure with preserved ejection fraction in patients with concurrent hypertension and diabetes. | At baseline
  Phenotypes of heart failure with preserved ejection fraction in patients with concurrent hypertension and diabetes.
Composite primary endpoint | 12 months - Up to 18 months from baseline
  Composite primary endpoint: Time to first event of composite outcome (all-cause mortality, or hospitalization for heart failure (HHF)) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
Combined endpoint | 12 months - Up to 18 months from baseline
  Combined endpoint: Time to first event of composite outcome (Cardiovascular mortality, or hospitalization for heart failure (HHF)) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and composite primary endpoint | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and composite primary endpoint: Time to first event of all-cause mortality, hospitalization for heart failure (HHF) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and combined endpoint | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and combined endpoint: Time to first event of CV mortality, hospitalization for heart failure (HHF) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.

SECONDARY OUTCOMES:
Occurence of HHF (first and recurrent) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  Occurence of HHF (first and recurrent) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
All cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  All cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
Cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  All cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
Time to first occurence of HHF (first and recurrent) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  Time to first occurence of HHF (first and recurrent) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
Time to first all cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes | 12 months- Up to 18 months from baseline
  Time to first all cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes
Time to first cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  Time to first cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.

OTHER OUTCOMES:
The correlation between clinical phenotypes and time to the first occurence of HHF (first and recurrent) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and time to the first occurence of HHF (first and recurrent) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and time to all cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and time to all cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and time to cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and time to cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and the occurence of HHF (first and recurrent) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and the occurence of HHF (first and recurrent) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and all cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and all cause mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and combined endpoint of cardiovascular mortality and cardiovascular hospitalization in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and combined endpoint of cardiovascular mortality and cardiovascular hospitalization in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and non-cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and non- cardiovascular mortality in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between clinical phenotypes and non-cardiovascular hospitalization in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes. | 12 months- Up to 18 months from baseline
  The correlation between clinical phenotypes and non- cardiovascular hospitalization in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
Risk stratification of HFpEF in patients with hypertension and diabetes using the echocardiographic and natriuretic peptide score from the HFA-PEFF algorithm. | At baseline
  Risk stratification of heart failure with preserved ejection fraction in patients with hypertension and diabetes using the echocardiographic and natriuretic peptide score from the HFA-PEFF (Heart Failure Association- Pretest, Echocardiogaphic and Natriuretic peptide score, Functional testing and Final etiology) algorithm. This score ranges from 0 to 6, with higher score predicts worse outcome.
Risk stratification of heart failure with preserved ejection fraction in patients with hypertension and diabetes using the H2FPEF (Heavy, Hypertension, atrial Fibrillation, Pulmonary hypertension, Elder, Filling pressure) score. | At baseline
  Risk stratification of heart failure with preserved ejection fraction in patients with hypertension and diabetes using the H2FPEF (Heavy, Hypertension, atrial Fibrillation, Pulmonary hypertension, Elder, Filling pressure) score. Maximum score is 9, minimum is 0. Higher score predicts worse outcome.
The correlation between echocardiographic and natriuretic peptide score from the HFA-PEFF algorithm and time to composite endpoint (all-cause mortality or HHF) | 12 months- Up to 18 months from baseline
  The correlation between echocardiographic and natriuretic peptide score from the HFA-PEFF (Heart Failure Association- Pretest, Echocardiographic and Natriuretic peptide score, Functional testing and Final etiology) algorithm and time to composite endpoint (all-cause mortality and HHF) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
The correlation between H2FPEF (Heavy, Hypertension, atrial Fibrillation, Pulmonary hypertension, Elder, Filling pressure) score and time to composite endpoint (all-cause mortality and HHF) | 12 months- Up to 18 months from baseline
  The correlation between H2FPEF score (Heavy, Hypertension, atrial Fibrillation, Pulmonary hypertension, Elder, Filling pressure) and time to composite endpoint (all-cause mortality and HHF) in patients with heart failure with preserved ejection fraction and concurrent hypertension, diabetes.
Comparing diagnostic criteria for heart failure with preserved ejection fraction using 2016 ESC guideline, HFA-PEFF score and H2FPEF score in patients with hypertension and diabetes. | At baseline
  Comparing diagnostic criteria for heart failure with preserved ejection fraction using 2016 ESC (European Society of Cardiology) guideline, HFA-PEFF (Heart Failure Association- Pretest, Echocardiographic and Natriuretic peptide score, Functional testing and Final etiology) algorithm and H2FPEF (Heavy, Hypertension, atrial Fibrillation, Pulmonary hypertension, Elder, Filling pressure) score in patients with hypertension and diabetes.
The prevalence of undiagnosed heart failure with preserved ejection fraction in patients with hypertension and diabetes presenting with signs and symptoms of heart failure. | At baseline
  The prevalence of undiagnosed heart failure with preserved ejection fraction in patients with hypertension and diabetes presenting with signs and symptoms of heart failure.
The prevalence of chronic kidney disease, persistent albuminuria, coronary artery disease, atrial fibrillation, and anemia in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes | At baseline
  The prevalence of chronic kidney disease, persistent albuminuria, coronary artery disease, atrial fibrillation, and anemia in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes
The incidence of chronic kidney disease, persistent albuminuria, coronary artery disease, atrial fibrillation and anemia in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes | 12 months- Up to 18 months from baseline
  The incidence of chronic kidney disease, persistent albuminuria, coronary artery disease, atrial fibrillation and anemia in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes
The correlation between baseline chronic kidney disease, persistent albuminuria, coronary artery disease, atrial fibrillation, anemia and mortality in patients with diabetes, hypertension and heart failure with preserved ejection fraction | 12 months- Up to 18 months from baseline
  The correlation between baseline chronic kidney disease, persistent albuminuria, coronary artery disease, atrial fibrillation, anemia and mortality in patients with diabetes, hypertension and heart failure with preserved ejection fraction
Change in ejection fraction overtime in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes | 12 months- Up to 18 months from baseline
  Change in ejection fraction overtime in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes
Change in structural abnormality on echocardiogram overtime in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes | 12 months- Up to 18 months from baseline
  Change in structural abnormality on echocardiogram overtime in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes
Change in severity of diastolic dysfunction overtime in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes | 12 months- Up to 18 months from baseline
  Change in severity of diastolic dysfunction overtime in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes
The correlation between baseline level of NT-proBNP and composite endpoint (all-cause mortality and HHF) in patients with diabetes, hypertension and heart failure with preserved ejection fraction | 12 months- Up to 18 months from baseline
  The correlation between baseline level of NT-proBNP and composite endpoint (all-cause mortality and HHF) in patients with diabetes, hypertension and heart failure with preserved ejection fraction
The correlation between change in NT-proBNP level overtime and composite endpoint (all-cause mortality and HHF) in patients with diabetes, hypertension and heart failure with preserved ejection fraction | 12 months- Up to 18 months from baseline
  The correlation between change in NT-proBNP level overtime and composite endpoint (all-cause mortality and HHF) in patients with diabetes, hypertension and heart failure with preserved ejection fraction
Change in eGFR overtime in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes | 12 months- Up to 18 months from baseline
  Change in eGFR overtime in patients with heart failure with preserved ejection fraction and concurrent hypertension and diabetes
Simultaneous risk factor control (HbA1c (%), and LDL-c (mmol/L), and blood pressure (mmHg)) in patients with diabetes, hypertension and heart failure with preserved ejection fraction | 12 months- Up to 18 months from baseline
  Simultaneous risk factor control (HbA1c (%), and LDL-c (mmol/L), and blood pressure (mmHg)) in patients with diabetes, hypertension and heart failure with preserved ejection fraction
Change in simultaneous risk factor control (HbA1c (%), and LDL-c (mmol/L), and blood pressure (mmHg)) overtime in patients with diabetes, hypertension and heart failure with preserved ejection fraction | 12 months- Up to 18 months from baseline
  Change in simultaneous risk factor control (HbA1c (%), and LDL-c (mmol/L), and blood pressure (mmHg)) in patients with diabetes, hypertension and heart failure with preserved ejection fraction
The correlation between simultaneous risk factor control and composite endpoint (all-cause mortality and HHF) in patients with diabetes, hypertension and heart failure with preserved ejection fraction | 12 months- Up to 18 months from baseline
  The correlation between simultaneous risk factor control and composite endpoint (all-cause mortality and HHF) in patients with diabetes, hypertension and heart failure with preserved ejection fraction
The correlation between simultaneous risk factor control (HbA1c (%), and LDL-c (mmol/L), and blood pressure (mmHg)) and mortality in patients with diabetes, hypertension and heart failure with preserved ejection fraction | 12 months- Up to 18 months from baseline
  The correlation between simultaneous risk factor control (HbA1c (%), and LDL-c (mmol/L), and blood pressure (mmHg)) and mortality in patients with diabetes, hypertension and heart failure with preserved ejection fraction

CONTACTS AND LOCATIONS:
Overall Officials: Van Ngoc-Thanh Nguyen, MD, MSci, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (2):
- Vietnam (2):
  - Nhan Dan Gia Dinh Hospital, Ho Chi Minh City, Ho Chi Minh
  - University Medical Center, Ho Chi Minh City